CLINICAL TRIAL: NCT04558359
Title: Renin and Renal Biomarker Response to Angiotensin II Versus Controls in Septic Shock: An Open-Label Study
Brief Title: Renin and Renal Biomarker Response to Angiotensin II
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alexander Flannery (Other)
Responsible Party: Sponsor-Investigator, Alexander Flannery, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 57411
Record Dates: First submitted 2020-09-07; First posted 2020-09-22 (Actual); Results first posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Septic Shock; Acute Kidney Injury
Keywords: Renin; Angiotensin II; vasopressor; sepsis
MeSH Terms: conditions — Shock, Septic; Acute Kidney Injury; Sepsis | interventions — Standard of Care; Angiotensin II

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard of Care Cohort (Active Comparator): Patients in this group will receive standard of care treatment.
  Interventions: Other: Standard of Care
- Angiotensin II Cohort (Experimental): Patients in this group will receive angiotensin II.
  Interventions: Drug: Angiotensin II

INTERVENTIONS:
Other: Standard of Care — These patients will receive standard of care treatment. Plasma renin levels and biomarkers of renal function will be measured.
  Arms: Standard of Care Cohort
Drug: Angiotensin II — These patients will receive angiotensin II in addition to standard of care treatment. Plasma renin levels and biomarkers of renal function will be measured.
  Arms: Angiotensin II Cohort

SUMMARY:
Septic shock continues to exert a large economic burden around the world. Several developments have occurred that lead to the current study. First, angiotensin II is the newest FDA approved vasopressor agent indicated for use in vasodilatory shock. Several subgroups from the approval trial have indicated that angiotensin II may confer a survival benefit in certain conditions, including those patients requiring continuous renal replacement therapy, those with altered angiotensin I: angiotensin II ratios, and most recently, those with elevated renin levels (which may serve as a surrogate for dysfunctional angiotensin 1: angiotensin II ratios). This open-label, sequential period pilot study will evaluate angiotensin II and biomarker response (renin) in the treatment of septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Medical ICU admission
* Septic shock
* Norepinephrine requirement = 0.15 mcg/kg/min for = 30 minutes (if cirrhosis, norepinephrine requirement = 0.1 mcg/kg/min for = 30 minutes)
* Kidney Disease Improving Global Outcomes stage 1 or greater Acute Kidney Injury

Exclusion Criteria:

* Prisoner
* Pregnancy
* Acute occlusive coronary syndrome requiring intervention or acute myocardial infarction of any degree
* Purely cardiogenic shock (no distributive component)
* Mesenteric ischemia
* Acute ischemic stroke
* Hemorrhagic shock
* Active treatment of hepatorenal syndrome targeting a Mean Arterial Pressure = 65 mm Hg
* Planned withdrawal of care within next 24 hours or no escalation of care
* Patient enrolled in an interventional study
* High likelihood of medical futility in using this drug:
* 3 or more vasopressors required to sustain MAP
* Sustained norepinephrine equivalents > 0.5 mcg/kg/min
* COVID-19 positive, or high suspicion of COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2023-07-24 (Actual); Study Completion 2023-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander H Flannery, Pharm.D., Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky HealthCare Chandler Medical Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 enrolled participants in the angiotensin II arm had changes in status that deemed them ineligible for the study and they subsequently did not receive open label angiotensin II.
Period: Overall Study
Arm/Group | Standard of Care Cohort | Angiotensin II Cohort
Started | 10 | 18
Completed | 10 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care Cohort | Angiotensin II Cohort | Total
Number analyzed (Participants) | 10 | 18 | 28
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63 [53 to 66] | 61 [48 to 69] | 62 [50 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 5 | 11 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 9 | 16 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 18 | 28

OUTCOME MEASURES:

1. Primary Outcome: Change in Plasma Renin Levels
Description: Plasma renin levels will be measured from blood collected at baseline, 24 hours, and at shock resolution. Additionally, a 3-hour measurement will be included in the angiotensin II arm.
Time Frame: Until shock resolution, up to 14 days (at baseline, 3 hours, 24 hours, and shock resolution, up to 14 days)
Population: Number analyzed in one or more rows may be different from overall number due to participant death which would preclude subsequent measurements. 3-hour sample was only done in the angiotensin II arm.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Standard of Care Cohort | Angiotensin II Cohort
Number analyzed (Participants) | 10 | 18
pg/mL
  Baseline Minus 24-Hour Sample: number analyzed (Participants) | 7 | 18
  Baseline Minus 24-Hour Sample | -15 [-291 to 38] | 69 [1 to 352]
  Baseline Minus Shock Resolution: number analyzed (Participants) | 6 | 11
  Baseline Minus Shock Resolution | -6 [-101 to 372] | 26 [13 to 340]
  Baseline Minus 3-Hour: number analyzed (Participants) | 0 | 18
  Baseline Minus 3-Hour |  | 41 [1 to 292]

2. Secondary Outcome: Change in Plasma Cystatin C
Description: Cystatin C will be measured from blood collected at baseline, 24 hours, and at shock resolution.
Time Frame: Until shock resolution, up to 14 days (at baseline, 3 hours, 24 hours, and shock resolution, up to 14 days)
Population: Number analyzed in one or more rows may be different from overall number due to participant death which would preclude subsequent measurements. 3-hour sample was done only in the angiotensin II arm.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Standard of Care Cohort | Angiotensin II Cohort
Number analyzed (Participants) | 10 | 18
ng/mL
  Baseline Minus 24-Hour: number analyzed (Participants) | 7 | 18
  Baseline Minus 24-Hour | -254 [-731 to 932] | -143 [-762 to 121]
  Baseline Minus Shock Resolution: number analyzed (Participants) | 6 | 11
  Baseline Minus Shock Resolution | 99 [-920 to 815] | -124 [-524 to 644]
  Baseline Minus 3-Hour: number analyzed (Participants) | 0 | 18
  Baseline Minus 3-Hour |  | -196 [-527 to 329]

3. Secondary Outcome: Days to Discontinuation of Catecholamines
Description: Days from enrollment to discontinuation of catecholamines
Time Frame: Until shock resolution, up to 14 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Standard of Care Cohort | Angiotensin II Cohort
Number analyzed (Participants) | 10 | 18
days | 0.9 [0.5 to 3.2] | 3.5 [1.3 to 6.4]

4. Secondary Outcome: ICU Length of Stay
Description: Number of days in the intensive care unit (ICU).
Time Frame: From enrollment to ICU discharge, up to 28 days following enrollment
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Standard of Care Cohort | Angiotensin II Cohort
Number analyzed (Participants) | 10 | 18
days | 4.3 [1.0 to 8.5] | 7.2 [3.0 to 11.5]

5. Secondary Outcome: Number of Participants With In-hospital Mortality
Description: Assessment of all-cause mortality within hospital admission
Time Frame: Up to 3 months following enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Cohort | Angiotensin II Cohort
Number analyzed (Participants) | 10 | 18
Participants | 9 | 9

6. Secondary Outcome: Renal Replacement Therapy-free Days
Description: Days free of renal replacement therapy from enrollment up to day 28
Time Frame: Within 28 days of enrollment
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Standard of Care Cohort | Angiotensin II Cohort
Number analyzed (Participants) | 10 | 18
days | 0 [0 to 0] | 21 [0 to 28]

7. Secondary Outcome: Number of Participants Experiencing Prespecified Safety Outcomes
Description: Incidence of venous thromboembolism, arrhythmia, extremity hypoperfusion, delirium, new ischemic event, new infection
Time Frame: Up to 72 hours following shock resolution, no longer than 17 days from enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Cohort | Angiotensin II Cohort
Number analyzed (Participants) | 10 | 18
Participants | 0 | 0

8. Secondary Outcome: Change in Plasma Neutrophil Gelatinase-associated Lipocalin (NGAL)
Description: NGAL will be measured from blood collected at baseline, 24 hours, and at shock resolution.
Time Frame: Until shock resolution, up to 14 days (at baseline, 3 hours, 24 hours, and shock resolution, up to 14 days)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Standard of Care Cohort | Angiotensin II Cohort
Number analyzed (Participants) | 10 | 18
ng/mL
  Baseline Minus 24-Hour: number analyzed (Participants) | 7 | 18
  Baseline Minus 24-Hour | 10 [-13 to 213] | 93 [-39 to 235]
  Baseline Minus Shock Resolution: number analyzed (Participants) | 6 | 11
  Baseline Minus Shock Resolution | 18 [-39 to 819] | 201 [66 to 421]
  Baseline Minus 3-Hour: number analyzed (Participants) | 0 | 18
  Baseline Minus 3-Hour |  | -21 [-75 to 85]

ADVERSE EVENTS:
Time Frame: Up to 72 hours following shock resolution, no longer than 17 days from enrollment
Description: Targeted screening for venous thromboembolism, arrhythmia, extremity hypoperfusion, delirium, new ischemic event, new infection from enrollment up to 72 hours following shock resolution.
Arm/Group | Standard of Care Cohort | Angiotensin II Cohort
All-Cause Mortality (participants affected / at risk) | 9/10 | 9/18
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/18
Other Adverse Events (participants affected / at risk) | 0/10 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-19): https://cdn.clinicaltrials.gov/large-docs/59/NCT04558359/Prot_SAP_000.pdf